CLINICAL TRIAL: NCT00678327
Title: A Randomized Phase III Trial to Assess Response Adapted Therapy Using FDG-PET Imaging in Patients With Newly Diagnosed, Advanced Hodgkin Lymphoma
Brief Title: Fludeoxyglucose F 18-PET/CT Imaging in Assessing Response to Chemotherapy in Patients With Newly Diagnosed Stage II, Stage III, or Stage IV Hodgkin Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other); Cancer Research UK & UCL Cancer Trials Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000593562; CRUK-2007-006064-30; CRUK-07/146
Record Dates: First submitted 2008-05-09; First posted 2008-05-15 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; adult nodular sclerosis Hodgkin lymphoma; adult lymphocyte depletion Hodgkin lymphoma; adult lymphocyte predominant Hodgkin lymphoma; adult mixed cellularity Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Filgrastim; pegfilgrastim; Cyclophosphamide; Dacarbazine; Doxorubicin; Etoposide; Prednisolone; Procarbazine; Vinblastine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Active Comparator): Patients receive ABVD chemotherapy comprising doxorubicin hydrochloride IV, bleomycin IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bleomycin sulfate; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine sulfate
- Arm II (Active Comparator): Patients receive AVD chemotherapy comprising doxorubicin hydrochloride IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: vinblastine sulfate
- BEACOPP-14 chemotherapy (Experimental): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; etoposide IV on days 1-3; oral procarbazine hydrochloride and oral prednisolone on days 1-7; and bleomycin IV and vincristine IV on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 8-13 OR pegfilgrastim SC once on day 8. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisolone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate
- BEACOPP-escalated chemotherapy (Experimental): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; etoposide IV on days 1-3; oral procarbazine hydrochloride on days 1-7; oral prednisolone on days 1-14; and bleomycin IV and vincristine IV on day 8. Patients also receive G-CSF SC beginning on day 8 and continuing until blood counts recover OR pegfilgrastim SC once on day 8. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisolone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV
  Arms: Arm I; BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Biological: filgrastim — Given subcutaneously
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Biological: pegfilgrastim — Given subcutaneously
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Drug: cyclophosphamide — Given IV
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Drug: dacarbazine — Given IV
  Arms: Arm I; Arm II
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide — Given IV
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Drug: prednisolone — Given orally
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Drug: procarbazine hydrochloride — Given orally
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy
Drug: vinblastine sulfate — Given IV
  Arms: Arm I; Arm II
Drug: vincristine sulfate — Given IV
  Arms: BEACOPP-14 chemotherapy; BEACOPP-escalated chemotherapy

SUMMARY:
RATIONALE: Imaging procedures, such as fludeoxyglucose F 18 (FDG)-PET/CT scan, done before, during, and after chemotherapy may help doctors assess a patient's response to treatment and help plan the best treatment. It is not yet known whether FDG-PET/CT imaging is effective in assessing response to chemotherapy in patients with newly diagnosed Hodgkin lymphoma.

PURPOSE: This randomized phase III trial is studying FDG-PET/CT imaging to see how well it works in assessing response to chemotherapy in patients with newly diagnosed stage II, stage III, or stage IV Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if fludeoxyglucose F 18 (FDG)-PET/CT imaging can be reproducibly and effectively applied in the early assessment of response to chemotherapy in patients with newly diagnosed stage II-IV Hodgkin lymphoma.
* To determine if a negative FDG-PET/CT scan after 2 courses of ABVD chemotherapy comprising doxorubicin hydrochloride, bleomycin, vinblastine, and dacarbazine can be used to predict a group of patients for whom it is safe to reduce therapy by the subsequent omission of bleomycin, without detriment to progression-free survival.
* To determine if treatment intensification in response to positive FDG-PET/CT imaging after 2 courses of ABVD chemotherapy can improve the outcome by comparison with previous series.

OUTLINE: This is a multicenter study.

Patients undergo fludeoxyglucose F 18 (FDG)-PET/CT imaging at baseline. Patients then receive ABVD chemotherapy comprising doxorubicin hydrochloride IV, bleomycin IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Between days 22 and 25 of course 2, patients undergo a second FDG-PET/CT scan to assess response. Subsequent therapy is based on FDG-PET/CT scan results.

* Negative FDG-PET/CT scan: Patients with a negative FDG-PET/CT scan are randomized to 1 of 2 treatment arms.

  * Arm I (ABVD chemotherapy): Patients receive ABVD chemotherapy comprising doxorubicin hydrochloride IV, bleomycin IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II (AVD chemotherapy): Patients receive AVD chemotherapy comprising doxorubicin hydrochloride IV, vinblastine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
* Positive FDG-PET/CT scan: Patients with a positive FDG-PET/CT scan are assigned to 1 of 2 chemotherapy regimens, as determined by the participating center.

  * BEACOPP-14 chemotherapy: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; etoposide IV on days 1-3; oral procarbazine hydrochloride and oral prednisolone on days 1-7; and bleomycin IV and vincristine IV on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 8-13 OR pegfilgrastim SC once on day 8. Treatment repeats every 14 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * BEACOPP-escalated chemotherapy: Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV on day 1; etoposide IV on days 1-3; oral procarbazine hydrochloride on days 1-7; oral prednisolone on days 1-14; and bleomycin IV and vincristine IV on day 8. Patients also receive G-CSF SC beginning on day 8 and continuing until blood counts recover OR pegfilgrastim SC once on day 8. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of BEACOPP chemotherapy, patients undergo a third FDG-PET/CT scan to assess response. Patients with a negative FDG-PET/CT scan receive 2 more courses of BEACOPP-14 or 1 more course of BEACOPP-escalated chemotherapy. Patients with a persistently positive FDG-PET/CT scan may receive radiotherapy to sites of FDG uptake or salvage chemotherapy, at the investigator's discretion.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin lymphoma (HL) meeting the following criteria:

  * Meets current WHO classification criteria (i.e., nodular sclerosis, mixed cellularity, lymphocyte rich, and lymphocyte-depleted)
  * Clinical stage IIB, III, or IV disease OR clinical stage IIA disease with adverse features, including any of the following:

    * Bulk mediastinal disease, defined as maximal transverse diameter of mass > 0.33 of the internal thoracic diameter at D5/6 interspace on routine chest x-ray
    * Disease outside the mediastinum and lymph node or lymph node mass > 10 cm in diameter
    * More than two sites of disease
    * Other poor-risk features that require treatment with full course combination chemotherapy
* Newly diagnosed disease
* No CNS or meningeal involvement by lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 3 months
* ANC > 1,500/mm^3 (unless there is bone marrow infiltration by lymphoma)
* Platelet count > 100,000/mm^3 (unless there is bone marrow infiltration by lymphoma)
* Creatinine < 150% of upper limit of normal (ULN)
* Bilirubin < 2.0 times ULN (unless attributed to lymphoma)
* Transaminases < 2.5 times ULN (unless attributed to lymphoma)
* LVEF ≥ 50% (in patients with a significant history of ischemic heart disease or hypertension)
* Diffusion capacity within 25% of normal predicted value by lung function testing
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Amenable to the administration of a full course of chemotherapy, according to the investigator
* Must have access to PET/CT scanning
* No poorly controlled diabetes mellitus
* No cardiac contraindication to doxorubicin hydrochloride, including abnormal contractility by ECHO or MUGA
* No neurological contraindication to chemotherapy (e.g., pre-existing neuropathy)
* No other concurrent uncontrolled medical condition
* No other active malignant disease within the past 10 years, except fully excised basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix
* No known positivity for HIV, hepatitis B surface antigen, or hepatitis C

  * Routine testing, in the absence of risk factors, is not required
* No medical or psychiatric condition that compromises the patient's ability to give informed consent

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy or other investigational drug for HL

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1202 (Actual)
Dates: Start 2008-08-29 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
3-year progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years after last patient recruited
Acute and chronic toxicity as assessed by NCI CTCAE v3.0 | 5 years after last patient recruited

CONTACTS AND LOCATIONS:
Overall Officials: Peter Johnson, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southampton, England, United Kingdom

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Luminari S, Fossa A, Trotman J, Molin D, d'Amore F, Enblad G, Berkahn L, Barrington SF, Radford J, Federico M, Kirkwood AA, Johnson PWM. Long-Term Follow-Up of the Response-Adjusted Therapy for Advanced Hodgkin Lymphoma Trial. J Clin Oncol. 2024 Jan 1;42(1):13-18. doi: 10.1200/JCO.23.01177. Epub 2023 Oct 26. PMID 37883739
- [Derived] Anderson RA, Remedios R, Kirkwood AA, Patrick P, Stevens L, Clifton-Hadley L, Roberts T, Hatton C, Kalakonda N, Milligan DW, McKay P, Rowntree C, Scott FM, Johnson PWM. Determinants of ovarian function after response-adapted therapy in patients with advanced Hodgkin's lymphoma (RATHL): a secondary analysis of a randomised phase 3 trial. Lancet Oncol. 2018 Oct;19(10):1328-1337. doi: 10.1016/S1470-2045(18)30500-X. Epub 2018 Sep 13. PMID 30220622
- [Derived] Johnson P, Federico M, Kirkwood A, Fossa A, Berkahn L, Carella A, d'Amore F, Enblad G, Franceschetto A, Fulham M, Luminari S, O'Doherty M, Patrick P, Roberts T, Sidra G, Stevens L, Smith P, Trotman J, Viney Z, Radford J, Barrington S. Adapted Treatment Guided by Interim PET-CT Scan in Advanced Hodgkin's Lymphoma. N Engl J Med. 2016 Jun 23;374(25):2419-29. doi: 10.1056/NEJMoa1510093. PMID 27332902